CLINICAL TRIAL: NCT02009319
Title: Endobronchial Ultrasound Elastography: the Utility of Strain Ratio for Lymph Node Staging in Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Principal Investigator, Aleš Rozman, MD, specialist from pulmonary diseases, The University Clinic of Pulmonary and Allergic Diseases Golnik
Other Study IDs: ENDO - 004
Record Dates: First submitted 2013-12-04; First posted 2013-12-12 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Lung Cancer
Keywords: endobronchial ultrasound; EBUS - TBNA; elastography; strain ratio; lung cancer staging
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EBUS TBNA lymph node specimen - a part of routine diagnostic procedure
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this pilot study is to evaluate EBUS elastography strain ratio in assessment of mediastinal lymph nodes in patients with suspicion for lung cancer for the first time. Strain ratios of mediastinal lymph nodes will be compared with EBUS B-mode features and with tissue diagnosis as a gold standard.

DETAILED DESCRIPTION:
Evaluation will be performed on consenting consecutive patients at least 18 years old, referred to bronchoscopy with suspicion for lung cancer according to chest CT-scan. Eligible patients should have either enlarged discrete N2/N3 lymph nodes, or central tumor or enlarged N1 lymph nodes with normal mediastinal lymph nodes. Exclusion criteria will be metastatic disease, severe co-morbidity that disqualified surgical treatment, mediastinal infiltration by tumor and small peripheral lung tumor with normal-sized mediastinal lymph nodes.

Outcomes: Sensitivity, specificity, accuracy, positive predictive value (PPV) and negative predictive value (NPV) for probability of malignant lymph node diagnosis, determined by elastography strain ratio. Receiver operating characteristic (ROC) analysis will be made to display specificity / sensitivity for different strain ratio cut-off values. Area under the ROC curve will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* enlarged discrete N2/N3 lymph nodes
* central tumor with normal mediastinal lymph nodes
* enlarged N1 lymph nodes with normal mediastinal lymph nodes

Exclusion Criteria:

* metastatic disease
* severe co-morbidity that disqualified surgical treatment
* mediastinal infiltration by tumor
* small peripheral lung tumor with normal-sized mediastinal lymph nodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients at least 18 years old, referred to bronchoscopy with suspicion for lung cancer according to chest CT-scan
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
elastography strain ratio | up to 7 months
  Sensitivity, specificity, accuracy, positive predictive value (PPV) and negative predictive value (NPV)

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Pulmonary and Allergic Diseases Golnik, Golnik, Golnik, Slovenia